CLINICAL TRIAL: NCT06449027
Title: A Phase III, Multicenter, Randomized, Open-Label Study to Assess the Safety, Efficacy and Pharmacokinetic Behavior of Leuprolide Injectable Emulsion for Premenopausal Breast Cancer Subjects.
Brief Title: Safety, Efficacy and Pharmacokinetic Behavior of Leuprolide Injectable Emulsion for Premenopausal Breast Cancer Subjects.
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GenSci093-301
Record Dates: First submitted 2024-05-31; First posted 2024-06-07 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Subjects
MeSH Terms: interventions — Tamoxifen; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Leuprolide Injectable Emulsion (Experimental): 100 subjects were injected Leuprolide Injectable Emulsion 42mg every 24 weeks for 48 weeks.
  Interventions: Drug: T Leuprolide Injectable Emulsion
- Leuprorelin Acetate Microspheres for Injection (Active Comparator): 100 subjects were injected Leuprorelin Acetate Microspheres for Injection 11.25mg every 12 weeks for 48 weeks.
  Interventions: Drug: Leuprorelin Acetate Microspheres for Injection

INTERVENTIONS:
Drug: T Leuprolide Injectable Emulsion — Arm 1 subjects were injected Leuprolide Injectable Emulsion 42mg every 24 weeks for 48 weeks, and taked Tamoxifen Citrate Tablets 10mg bid for 48 weeks.
  Other Names: Tamoxifen Citrate Tablets
  Arms: Leuprolide Injectable Emulsion
Drug: Leuprorelin Acetate Microspheres for Injection — Arm 2 subjects were injected Leuprorelin Acetate Microspheres for Injection 11.25mg every 12 weeks for 48 weeks, and taked Tamoxifen Citrate Tablets 10mg bid for 48 weeks.
  Other Names: Tamoxifen Citrate Tablets
  Arms: Leuprorelin Acetate Microspheres for Injection

SUMMARY:
The study is to assess the safety, efficacy and pharmacokinetic Behavior of Leuprolide Injectable Emulsion for Premenopausal Breast Cancer Subjects.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-Label , non-inferiority phase III study . All premenopausal women breast cancer subjects were randomly allocated to either the study group or control group in a 1:1 ratio. Furthermore, all subjects received tamoxifen citrate treatment throughout the entire duration of the study. The efficacy of maintaining serum E2 levels ≤30 pg/mL at 4-48 weeks post-treatment will be assessed in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal female subjects aged 18 to 55 years old.
* Histological or cytological confirmation of HR+，HER2- premenopausal breast cancer.
* Subjects have any breast cancer surgery before informing, and no clinical residual local regional lesions were found after the surgery.
* Life expectancy is not less than 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate function of major organs.

Exclusion Criteria:

* History of evidence of distant metastatic lesions;
* Subjects have the history of new adjuvant or adjuvant endocrine treatment for breast cancer ( Excluding subjects receiving tamoxifen citrate tablets treatment for less than 12 weeks before informing).
* Active hepatitis B, hepatitis C or HIV in screening.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 211 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Observe the proportion of subjects whose E2 levels remain at postmenopausal levels between 4 and 48 weeks after treatment, to assess the Efficacy of Leuprolide Injectable Emulsion for Premenopausal Breast Cancer Subject. | 48 weeks

SECONDARY OUTCOMES:
Observe the concentration of LH, FSH, E2 after treatment. | 48 weeks
Pharmacokinetic Parameter(AUC) | 48 weeks
Pharmacokinetic Parameter(Cmax) | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, Doctor, Principal Investigator — Fudan University; Zhimin Shao, Doctor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China